CLINICAL TRIAL: NCT04094961
Title: Phase I/II Study of Twice Weekly Ixazomib Plus Pomalidomide and Dexamethasone in Relapsed/or Refractory Multiple Myeloma
Brief Title: Ixazomib + Pomalidomide + Dexamethasone In MM
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Omar Nadeem, MD (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Omar Nadeem, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-291
Record Dates: First submitted 2019-09-10; First posted 2019-09-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse
Keywords: Multiple Myeloma; Multiple Myeloma in Relapse
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ixazomib plus pomalidomide and dexamethasone (Experimental): The study drugs will be administered within a 21-day cycle
  * Phase I will follow a standard "3 +3" dose escalation design: Starting with the first cohort, 3 to 6 patients will be treated at this and each subsequent dose level.
  * The Phase II portion of the study will be a single-arm open-label enrollment with dosing based on the MTD determination in the Phase I portion of the study
  Interventions: Drug: Ixazomib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Oral, administered four times per cycle
  Other Names: Ninlaro®
Drug: Pomalidomide — Oral, administered 14 times per cycle
  Other Names: Pomalyst®
Drug: Dexamethasone — Oral, fixed dose administered 8 times per cycle
  Other Names: Baycadron; Decadron; Dexamethasone Intensol; DexPak; TaperDex; Zema-Pak; ZoDex; Zonacort

SUMMARY:
This is a Phase I/II study using the combination of twice weekly ixazomib plus pomalidomide and dexamethasone in relapsed and or refractory multiple myeloma (RRMM) patients.

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial. A Phase I clinical trial tests the safety of an investigational drug and tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA has approved both pomalidomide and ixazomib individually for the treatment of multiple myeloma. Dexamethasone, also FDA approved, is a type of steroid and is usually combined with other chemotherapy for the treatment of blood cancers, such as myeloma and leukemias.

* Ixazomib targets a part of cells called proteasomes. It works by slowing down or blocking proteasomes from doing their job of digesting proteins. In myeloma cells, there is a greater need for proteasomes to digest proteins; the buildup of excess proteins causes cell death.
* Pomalidomide has also been shown to cause tumor cell deaths. Dexamethasone can stop white blood cells from traveling to areas myeloma cells are causing damage. When combined with myeloma drugs, it sometimes makes those drugs work better.

In this research study, the investigators are:

* Testing the safety of ixazomib when given with pomalidomide and dexamethasone
* Pomalidomide and ixazomib are given individually for the treatment of multiple myeloma. Dexamethasone is also given for multiple myeloma
* Ixazomib when combined with pomalidomide and dexamethasone may help control the disease
* Ixazomib is FDA approved to treat multiple myeloma
* The investigators are looking for the highest dose of ixazomib that can be given safely in combination with pomalidomide and dexamethasone

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed and relapsed refractory myeloma may be eligible for this trial of they meet all the following entry criteria.
* Previously diagnosed with MM based on standard IMWG criteria and currently requires treatment.
* Patient has given voluntary written informed consent before performance of any study-related procedures not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care
* Patient had received at least two previous therapies OR received 1 prior line of therapy if previously treated with an IMiD plus a proteasome inhibitor and has demonstrated disease progression on or within 60 days of completion of the last therapy
* Patient has measurable disease defined as at least one of the following according to Standard Diagnostic Criteria (Rajkumar 2014):

  * Serum IgG, IgA, or IgM M-protein ≥ 0.5 g/dL, or
  * Serum IgD M-protein ≥ 0.05 g/dL, or
  * Urine M protein ≥200 mg/24 hours or
  * Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65)
  * Screening Laboratory evaluations within the following parameters

    * Absolute neutrophil count (ANC) ≥ 1,000 cells/dL (1.0 x 109/L) (Growth factors cannot be used more recently than 14 days prior to initiation of therapy)
    * Platelet count ≥ 75,000 cells/dL (75 x 109/L) (without transfusions required during the 14 days prior to initiation of therapy)
    * Hemoglobin ≥ 8.0 g/dl (RBC transfusions are permitted)
    * Total Bilirubin ≤ 1.5 X upper limit of normal (ULN) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
    * AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN
    * Calculated creatinine clearance ≥ 45 mL/min
  * ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
  * All study participants must be registered into the mandatory POMALYST REMS® program, and be willing and able to comply with the requirements of the POMALYST REMS® program.
  * Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the POMALYST REMS® program.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior exposure to ixazomib OR is refractory to pomalidomide
* Patients that have previously been treated with ixazomib, or participated in a study with ixazomib,whether treated with the agent or not, are also excluded
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
* Diagnosed or treated for another malignancy within 3 years prior to enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low risk prostate cancer after curative therapy.
* Known GI disease or is in need of, or has had a previous GI procedure that could interfere with the oral absorption or tolerance of ixazomib or pomalidomide including difficulty swallowing.
* Known central nervous system involvement.
* Systemic treatment, within 14 days before the first dose of treatment, with strong CYP3A or inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort OR systemic treatment within 14 days of the first dose of treatment with a strong inhibitor of CYP1A2 (ciprofloxacin, fluvoxamine, cimetidine, enoxacin, ethynyl estradiol, mexiletine)
* Any medical or psychiatric illness/social situation that in the Investigator's opinion, would impose excessive risk to the patient, would adversely affect his/her participating in this study or would limit compliance with study requirements.
* Any active, or uncontrolled cardiovascular conditions, including but not limited to uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, grade 3 thromboembolic event or myocardial infarction within the past 6 months.
* The following therapies within the stated time frames prior to initiation of therapy:

  * Previous cytotoxic therapies, including cytotoxic investigational agents, for multiple myeloma within 21 days (42 days for nitrosoureas).
  * The use of live vaccines within 30 days.
  * ImiDs or proteasome inhibitors within 14 days.
  * Other investigational therapies and/or monoclonal antibodies within 4 weeks.
  * Prior peripheral stem cell transplant within 12 weeks.
  * Prior allogeneic stem cell transplantation with active graft-versus-host-disease.
* Currently active graft versus host disease of any stage or grade after allogeneic stem cell transplantation
* Prior major surgical procedure or radiation therapy within 14 days of initiation of therapy.

  * Those who require a limited course of radiation for management of bone pain more than 14 days out from initiation of therapy are not excluded
  * If the involved field is small, 7 days will be considered a sufficient interval between radiotherapy and administration of the ixazomib.
* Daily requirement for corticosteroids (equivalent to > 10 mg/day prednisone, though >10mg/day is acceptable if physiological levels require, so long as the dose is stable for at least 7 days prior to initiation of therapy. Inhalation corticosteroids are exempt from this criterion.

  -- Lower amounts of corticosteroids that are not part of a daily requirement within 14 days prior to initiating therapy
* Concurrent symptomatic amyloidosis or plasma cell leukemia
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes)
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.

  -- Those who are on prophylactic antibiotics only, or on antibiotics and have confirmation of resolution of active infection are eligible.
* Known seropositive for active viral infection with human immunodeficiency virus (HIV) hepatitis B (HBV) or hepatitis C viral (HCV). Those who are seropositive because of hepatitis B vaccine are eligible. Patients who are positive for HBV core antibody or HBV surface antigen must have a negative polymerase chain reaction (PCR) result prior to enrollment. Those who are PCR positive will be excluded
* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Participants who are receiving any other investigational agents for any indication
* History of erythema multiforme or severe hypersensitivity to prior IMiD's® or those who have a known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Inability to tolerate thromboprophylaxis
* Failure to have fully recovered (≤ Grade 1 according to CTCAE v 5) from the reversible effects of prior chemotherapy
* Peripheral neuropathy must have resolved to Grade 1 toxicity or peripheral neuropathy grade 2 with no pain to be eligible
* Alopecia of any grade is eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity | 21 Days
  3 - 24 safety evaluable patients will be enrolled in up to 4 dose levels of ixazomib, pomalidomide and dexamethasone.
Overall Response Rate | 28 days
  Response will be evaluated using a Simon optimal two-stage design

SECONDARY OUTCOMES:
Time to Progression | time from first dose of study drug to progression, censored at date last known progression-free for those who have not progressed, whichever came first, assessed up to 60 months
  Estimated using the method of Kaplan-Meier.
Progression Free Survival | time from first dose of study drug to the disease progression or death from any cause, censored at date last known progression-free for those who have not progressed or died, whichever came first, assessed up to 60 months
  Estimated using the method of Kaplan-Meier.
Duration of Response | time from response to disease progression or death, or date last known progression-free and alive for those who have not progressed or died, whichever came first, assessed up to 60 months
  Estimated using the method of Kaplan-Meier.
Overall Survival | time from first dose of study drug to death or date last known alive, whichever came first, assessed up to 60 months
  Estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Nadeem, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: http://innovation@dfci.harvard.edu